CLINICAL TRIAL: NCT04109417
Title: Effect of Platelet-Rich Plasma Biomembrane on Enhancing Bone Regeneration Following Endodontic Surgery:A Prospective Randomized Clinical Trial
Brief Title: Effect of Platelet-Rich Plasma Biomembrane on Enhancing Bone Regeneration Following Endodontic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, salma genena, Lecturer of Endodontics, Conservative Dentistry Department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00010556
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteotomy filled with PRP-gel and covered with PRP-biomembrane (Experimental): the defect was filled with the previously activated autologous Platelet-rich plasma (PRP) gel and its supernatant. The site was then externally covered with the prepared bio-membrane composed of activated PRP which acted as an adjunct to the mucoperiosteal flap to stimulate tissue regeneration
  Interventions: Procedure: osteotomy filled with PRP-gel and covered with PRP-biomembrane
- osteotomy site left empty (Sham Comparator): osteotomy site following the surgical intervention was left empty
  Interventions: Procedure: osteotomy site following the surgical intervention was left empty

INTERVENTIONS:
Procedure: osteotomy filled with PRP-gel and covered with PRP-biomembrane
  Arms: osteotomy filled with PRP-gel and covered with PRP-biomembrane
Procedure: osteotomy site following the surgical intervention was left empty
  Arms: osteotomy site left empty

SUMMARY:
This study was conducted to evaluate clinical and radiographical outcome of using a standardized platelet-rich plasma (PRP) biomembrane following endodontic surgery and its correlation with the growth factors content in this concentrate.

DETAILED DESCRIPTION:
15 healthy patients of both genders, between 20 and 45 years of age, presenting with 22 anterior/premolar teeth in need of endodontic surgery were recruited. Teeth presented with failed non-surgical root canal therapy and periapical radiolucency of ≥ 1cm in size. Patients were randomly divided following surgery into two groups, with 11 teeth each.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients.
2. Selected tooth with previous root canal therapy failure and in need of endodontic surgery.
3. Existence of a periapical radiographic lesion surrounding the root canal treated tooth, of size ≥ 1 cm.
4. Healthy periodontal condition (probing depth, mobility & epithelial attachment level are all within normal range).

Exclusion Criteria:

1. Leaking coronal restoration.
2. Periodontal ligament breakdown and presence of apicomarginal defects.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
degree of periapical inflammation using periapical index (PAI) | baseline
  The PAI is a 5-point scale radiographic interpretation designed to determine the absence, presence, or transformation of a disease state. Each of the roots was categorized as: (1) Normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features. Each category used in the PAI represents a step on an ordinal scale of registration of periapical infection.
degree of periapical inflammation using periapical index (PAI) | 3 months
  The PAI is a 5-point scale radiographic interpretation designed to determine the absence, presence, or transformation of a disease state. Each of the roots was categorized as: (1) Normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features. Each category used in the PAI represents a step on an ordinal scale of registration of periapical infection.
degree of periapical inflammation using periapical index (PAI) | 6 months
  The PAI is a 5-point scale radiographic interpretation designed to determine the absence, presence, or transformation of a disease state. Each of the roots was categorized as: (1) Normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features. Each category used in the PAI represents a step on an ordinal scale of registration of periapical infection.
degree of periapical inflammation using periapical index (PAI) | 9 months
  The PAI is a 5-point scale radiographic interpretation designed to determine the absence, presence, or transformation of a disease state. Each of the roots was categorized as: (1) Normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features. Each category used in the PAI represents a step on an ordinal scale of registration of periapical infection.
degree of periapical inflammation using periapical index (PAI) | 12 months
  The PAI is a 5-point scale radiographic interpretation designed to determine the absence, presence, or transformation of a disease state. Each of the roots was categorized as: (1) Normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features. Each category used in the PAI represents a step on an ordinal scale of registration of periapical infection.
degree of periapical inflammation using periapical index (PAI) | 18 months
  The PAI is a 5-point scale radiographic interpretation designed to determine the absence, presence, or transformation of a disease state. Each of the roots was categorized as: (1) Normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features. Each category used in the PAI represents a step on an ordinal scale of registration of periapical infection.
degree of periapical inflammation using CBCT periapical index (CBCTPAI) | baseline
  CBCTPAI is a 6-point (0 -5) scoring system .The scores were calculated by analysis of the lesion in 3 dimensions, with CT slices being obtained in mesiodistal, buccopalatal, and diagonal directions. The score was determined by the largest extension of the lesion. The measurement of lesion depth in a CBCT image added the variables expansion of cortical bone (E) and destruction of cortical bone (D) usually detected starting from score 2.
degree of periapical inflammation using CBCT periapical index (CBCTPAI) | 18 months
  CBCTPAI is a 6-point (0 -5) scoring system .The scores were calculated by analysis of the lesion in 3 dimensions, with CT slices being obtained in mesiodistal, buccopalatal, and diagonal directions. The score was determined by the largest extension of the lesion. The measurement of lesion depth in a CBCT image added the variables expansion of cortical bone (E) and destruction of cortical bone (D) usually detected starting from score 2.
changes in bone mineral density of lesions in CBCT images | baseline
  region of interest measurements were made by the same operator in the sagittal view to provide consistency throughout the study protocol (baseline and at a 12 to 18 months post-operative interval). ROI was selected through drawing a polyline pattern that enabled us to include all the confines of the lesion (On Demand 3D® viewing software was used to obtain a mean grey level using the region of interest (ROI) polyline tool in sagittal plane images. The images of each CBCT scan were captured using the print screen button and exported into a Microsoft Word document as a record.
changes in bone mineral density of lesions in CBCT images | 18 months
  region of interest measurements were made by the same operator in the sagittal view to provide consistency throughout the study protocol (baseline and at a 12 to 18 months post-operative interval). ROI was selected through drawing a polyline pattern that enabled us to include all the confines of the lesion (On Demand 3D® viewing software was used to obtain a mean grey level using the region of interest (ROI) polyline tool in sagittal plane images. The images of each CBCT scan were captured using the print screen button and exported into a Microsoft Word document as a record.

SECONDARY OUTCOMES:
Platelet count in whole blood sample and in platelet rich plasma concentrate | baseline
  Platelet count in whole blood sample and in platelet rich plasma concentrate is assessed to detect fold increase in platelet count
concentration of Platelet-derived growth factor (PDGF) in the prepared PRP | baseline
  concentration of Platelet-derived growth factor (PDGF) in the prepared PRP was quantified using ELISA methods (R&D Center, Tokyo, Japan). The analyses were then performed as instructed by manufacturer
concentration of vascular endothelial growth factors (VEGF) in the prepared PRP | baseline
  Concentrations of VEGF growth factors in PRP was quantified using ELISA methods (R&D Center, Tokyo, Japan). The analyses were then performed as instructed by manufacturer

CONTACTS AND LOCATIONS:
Overall Officials: salma genena, PhD, Principal Investigator — Alexandria University
Locations (1):
- faculty of dentistry, Alexandria University, Alexandria, Egypt